CLINICAL TRIAL: NCT04588077
Title: Comparison the Seroconversion Rate Between Two-dose and Three-dose Regimens of Heplisav B Among Patients With Cirrhosis, a Randomized-control Prospective Study.
Brief Title: Comparison Between 2-dose Versus 3-dose Regimens of Heplisav B in Cirrhosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-24
Record Dates: First submitted 2020-09-18; First posted 2020-10-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B; Cirrhosis, Liver; Chronic Liver Disease
Keywords: hepatitis B vaccine; Heplisav-B; cirrhosis; chronic liver disease; 2 dose regimen; 3 dose regimen; non responder; poor responder; no response
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Fibrosis | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cirrhosis, 3-dose regimen (Experimental): Investigators will randomize the patient in the cirrhotic group to receive a 3-dose regimen of Heplisav-B.
  Interventions: Biological: Heplisav-B Injectable Product, 3-dose regimen
- Cirrhosis, 2-dose regimen (Active Comparator): Investigators will randomize the patient in the cirrhotic group to receive a 2-dose regimen of Heplisav-B.
  Interventions: Biological: Heplisav-B Injectable Product, 2-dose regimen
- Non cirrhosis, 3-dose regimen (Experimental): Investigators will randomize the patient in the noncirrhotic group to receive a 3-dose regimen of Heplisav-B.
  Interventions: Biological: Heplisav-B Injectable Product, 3-dose regimen
- Non cirrhosis, 2-dose regimen (Active Comparator): Investigators will randomize the patient in the noncirrhotic group to receive a 2-dose regimen of Heplisav-B.
  Interventions: Biological: Heplisav-B Injectable Product, 2-dose regimen

INTERVENTIONS:
Biological: Heplisav-B Injectable Product, 2-dose regimen — Investigators will randomly assign patients into a 2-dose regimen.
  Other Names: 2-dose regimen
  Arms: Cirrhosis, 2-dose regimen; Non cirrhosis, 2-dose regimen
Biological: Heplisav-B Injectable Product, 3-dose regimen — Investigators will randomly assign patients into a 3-dose regimen.
  Other Names: 3-dose regimen
  Arms: Cirrhosis, 3-dose regimen; Non cirrhosis, 3-dose regimen

SUMMARY:
Investigators want to compare the seroconversion rates between two-dose and three-dose regimens of the hepatitis B vaccine (Heplisav B) among patients with cirrhosis, a randomized prospective study.

DETAILED DESCRIPTION:
Study Rationale:

Hepatitis B virus is a major cause of acute and chronic liver disease both in the United States and worldwide. In 2016, an estimated 862,000 people were living with HBV infection in the US with a total of 1,649 U.S. death certificates recorded as an underlying or contributing cause of death. Chronic infection may cause liver cirrhosis and hepatocellular carcinoma (HCC). Since the introduction of the vaccine in the 1990s, there has been a significant decline in the incidence of HBV infection. Approved in November 2017, Heplisav-B uses a synthetic cytosine phosphoguanine oligonucleotide derived from bacterial DNA; it is thought to stimulate the immune system through activation of the toll-like receptor 9 pathway, which induces the production of cytokines such as interleukines such as interleukine-12 and interferon-alpha. It has been shown to induce higher immunity in healthy individuals compared to conventional vaccines.

The HBsAb titer should be checked 8 to 12 weeks after the administration of the vaccination series. Good responders were defined as those having the anti-HBs titer were ≥ 100 mUI/ml, poor responders having anti-HBs titer between 10 and 99 mUI/ml, and nonresponders having anti-HBs titer < 10 mIU/ml. The Seroprotection rate by age group in the healthy population is 100% in the 18-29-year-old group, 98.9% in the 30-29 %-year-old group, 97.2% in the 40-49-year-old group, 95.2% in the 50-59-year-old group, 91.6% in 60-70-year-old group. However, 5% of the general population will not mount a protection response.

Response to HBV vaccine is variable among patients with chronic diseases, such as HIV infection, celiac disease, IBD, end-stage renal disease, diabetes. The immunogenicity of the hepatitis B vaccine is also lower in decompensated cirrhosis. Among cirrhotic patients, only 45% who received Heplisav-B achieved immunity in investigator's previous retrospective analysis. The usual approach to HBV vaccine nonresponse is repeating the vaccine series in noninfected individuals.

Investigational Plan

*Study Design & Duration: Patients with cirrhosis or chronic liver disease presented to the hepatology clinic in Mercy Medical Center between 09/2020 and 07/2021 who do not have immunity against Hepatitis B (defined as anti-HBs titer < 10 mIU/ml) will be recruited. Patients will be stratified based on cirrhosis vs. no-cirrhosis and vaccine naive vs. vaccine experienced. Patients who had more than one vaccination series will not be included. Previous vaccination could be either Heplisav or Engerix; however, this information will be collected. The investigators' plan is to do the 1st part of the study is in treatment-naive patients and expand it to vaccine experienced.

Investigators will randomize patients to receive Heplisav-B in 0, 4 weeks, or Heplisav-B in 0, 4, 8 weeks. The HBV surface antibody titer will be checked 8 to 12 weeks after administration of the vaccination series and classified into good responders, poor responders, and nonresponders based on antibody titers.

Investigators will collect basic data including age, MELD scores, etiologies of cirrhosis (non-alcoholic fatty liver disease, hepatitis C, alcohol-induced liver disease, autoimmune liver disease, primary biliary cholangitis, primary sclerosing cholangitis, others), comorbidities (chronic obstructive pulmonary disease, diabetes mellitus, hypertension, coronary artery disease, renal failure, obesity), immunosuppressive drugs.

Primary endpoint: Seroconversion or immunity is defined as HBsAb level ≥ 10 mIU/ml.

Randomization process:

Investigators will use the envelope allocation technique. At first, Investigators will create a sequentially numbered random group assignment. The supplies for the randomization envelopes include envelopes, back carbon paper, and white copy paper. On the white copy paper, Investigators will write the study ID. Investigators will wrap the white copy paper inside the black carbon paper, put those into the envelope, and seal it.

The above data will be prospectively collected and entered into an excel database in a de-identified mode by giving them a coded number. Investigators will save data in a password-protected format and filed in the GI Research share drive and only the study staff will have access to the file to download for any study procedure or audit. It will be stored in a confidential manner, indefinitely in a secured Mercy share drive according to the 21 CFR part 11 guidelines.

The sample size for both arms: total 200. The current seroconversion rate of the hepatitis B vaccine in cirrhosis is low, about 50%, with the conventional schedule, either Engerix 0, 1 month, 6 months or Heplisav-B 0, 1 month. Investigators aim for the seroconversion rate of 70% with Heplisav-B 0, 1 month, 2 months. The probability of type I error is 5% and the power is 80%.

ELIGIBILITY:
Inclusion Criteria:

- All the cirrhosis patients more than 18 years old presented to the hepatology clinic in Mercy Medical Center between 09/2020 and 07/2021 who do not have immunity against Hepatitis B (defined as anti-HBs titer < 10 mIU/ml) will be recruited.

Exclusion Criteria:

* Anyone who has had a serious allergic reaction to a prior dose of the hepatitis B vaccine, a component of the hepatitis B vaccine, or yeast should not receive the hepatitis B vaccine.
* Those who had previous exposure to hepatitis B.
* Post liver transplant patients.
* Less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The rates of seroconversion after two doses of Heplisav-B given at 0 and 4 weeks versus three doses of Heplisav-B given at 0, 4 weeks, and 8 weeks. | 12 weeks after completing Heplisav-B series with two doses or three doses
  The rates of seroconversion is defined as an HBsAg antibody concentration ≥ 10 mIU/ml.

SECONDARY OUTCOMES:
Factors are associated with a lower likelihood of achieving immunogenicity, such as age, race, MELD scores, etiologies of cirrhosis, comorbidity, immunosuppressive drugs. Those information will be measured or described descriptively by chart review. | Through study completion, an average of 1 year
  Age (years) Race (White, Black, Other). MELD (Model For End-Stage Liver Disease) score: 6-40
  Etiologies of cirrhosis will include:
  Nonalcoholic Fatty Liver Disease (Yes/No). Hepatitis C (Yes/No). Alcohol induced Liver Disease (Yes/No). Autoimmune Hepatitis (Yes/No). Primary Biliary Cholangitis (Yes/No). Primary Sclerosing Cholangitis (Yes/No).
  Comorbidity will include:
  Chronic obstructive pulmonary disease (Yes/No). Diabetes mellitus (Yes/No). Hypertension (Yes/No). Coronary artery disease (Yes/No). Acute renal injury (Yes/No). Chronic renal disease (Yes/No). Obesity (Yes/No). The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared. A BMI of 30 and higher is considered obese. Immunosuppressive drugs (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Thuluvath, MD, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] A two-dose hepatitis B vaccine for adults (Heplisav-B). Med Lett Drugs Ther. 2018 Jan 29;60(1539):17-18. No abstract available. PMID 29364196
- [Result] Roni DA, Pathapati RM, Kumar AS, Nihal L, Sridhar K, Tumkur Rajashekar S. Safety and efficacy of hepatitis B vaccination in cirrhosis of liver. Adv Virol. 2013;2013:196704. doi: 10.1155/2013/196704. Epub 2013 Jun 6. PMID 23840211
- [Result] Jackson S, Lentino J, Kopp J, Murray L, Ellison W, Rhee M, Shockey G, Akella L, Erby K, Heyward WL, Janssen RS; HBV-23 Study Group. Immunogenicity of a two-dose investigational hepatitis B vaccine, HBsAg-1018, using a toll-like receptor 9 agonist adjuvant compared with a licensed hepatitis B vaccine in adults. Vaccine. 2018 Jan 29;36(5):668-674. doi: 10.1016/j.vaccine.2017.12.038. Epub 2017 Dec 27. PMID 29289383
- [Result] Yanny B, Konyn P, Najarian LM, Mitry A, Saab S. Management Approaches to Hepatitis B Virus Vaccination Nonresponse. Gastroenterol Hepatol (N Y). 2019 Feb;15(2):93-99. PMID 31011303
- [Result] Shetty A, Jun Yum J, Saab S. The Gastroenterologist's Guide to Preventive Management of Compensated Cirrhosis. Gastroenterol Hepatol (N Y). 2019 Aug;15(8):423-430. PMID 31592079
- [Result] Amjad W, Alukal J, Zhang T, Maheshwari A, Thuluvath PJ. Two-Dose Hepatitis B Vaccine (Heplisav-B) Results in Better Seroconversion Than Three-Dose Vaccine (Engerix-B) in Chronic Liver Disease. Dig Dis Sci. 2021 Jun;66(6):2101-2106. doi: 10.1007/s10620-020-06437-6. Epub 2020 Jul 2. PMID 32617767

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04588077/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04588077/ICF_000.pdf